CLINICAL TRIAL: NCT05194397
Title: Intensive Tailored Exercise Training With NAD+ Precursor Supplementation to Improve Muscle Mass and Fitness in Adolescent and Young Adult Hematopoietic Cell Transplant Survivors
Brief Title: Exercise Training and NR Supplementation Trial to Improve Fitness in AYA HCT Survivors
Acronym: IAMFIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); City of Hope Medical Center (Other); St. Jude Children's Research Hospital (Other); National Cancer Institute (NCI) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-017320; 1R01CA254955-01A1 (NIH)
Record Dates: First submitted 2021-12-09; First posted 2022-01-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Lymphoblastic Leukemia; Cancer Survivors; Aplastic Anemia; Myelodysplastic Syndromes; Myeloid Leukemia
Keywords: Sarcopenia; NAD+; Exercise Intervention; OXPHOS Capacity; VO2 Max; Adolescent young adults; Cancer Survivors; Hematopoietic Stem Cell Transplantation (HCT)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Aplastic; Myelodysplastic Syndromes; Leukemia, Myeloid; Sarcopenia | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled trial with a 2x2 factorial design testing the effects of an NAD+ precursor (NR) and exercise.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants and the investigator team will be blinded as to the group assignment: NR vs Placebo. All collected data (e.g., questionnaires) will be coded, so initial analysis will be conducted without knowledge of the participant's group status.
  While the assignment of participants to the exercise groups will not be blinded to the participant or majority of the study team, a designated blinded technician will perform the follow-up Cardio Pulmonary Exercise Testing. Follow-Up Cardio Pulmonary Exercise Testing will be performed by a dedicated blinded study team member, an exercise technician, who will not know if the participant was assigned to an arm including the exercise intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nicotinamide Riboside (NR) (Experimental): Investigators will use Good Manufacturing Process (GMP)-grade 300 mg capsules of the dietary supplement nicotinamide riboside (ChromaDex, Irvine CA). Investigators dose based on body weight, and monitor for adverse effects (AEs).
  For individuals with weight > 72 kg: 900 mg po qd x 16 wks.
  For individuals with weight > 48 kg and ≤ 72 kg: 600 mg po qd x 16 wks.
  For individuals with weight 24 ≤ 48 kg: 300 mg po qd x 16 wks.
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo (Placebo Comparator): Matched placebo will contain the same excipients without the active supplement and is generally recognized as safe. The placebo will be covered in an identical capsule (NR will be covered in the same capsule). Doses of placebo will match the body weight schema for dosing of NR. Investigators dose based on body weight, and monitor for adverse effects (AEs).
  For individuals with weight > 72 kg: 900 mg po qd x 16 wks.
  For individuals with weight > 48 kg and ≤ 72 kg: 600 mg po qd x 16 wks.
  For individuals with weight 24 ≤ 48 kg: 300 mg po qd x 16 wks.
  Interventions: Dietary Supplement: Placebo
- Exercise Intervention and NR (Experimental): The exercise program consists of at-home training sessions including: aerobic and strengthening components designed to progress persons gradually to 150-300 minutes of the equivalent of moderate aerobic activity, and twice weekly strength training exercises.
  Participants in this arm will receive both the Exercise Intervention and the NR.
  Interventions: Dietary Supplement: Nicotinamide Riboside; Other: Exercise Intervention
- Exercise Intervention and Placebo (Experimental): The exercise program consists of at-home training sessions including: aerobic and strengthening components designed to progress persons gradually to 150-300 minutes of the equivalent of moderate aerobic activity, and twice weekly strength training exercises.
  Participants in this arm will receive both the Exercise Intervention and the Placebo
  Interventions: Dietary Supplement: Placebo; Other: Exercise Intervention

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Investigators will use (Good Manufacturing Process) GMP-grade 300 mg capsules of the dietary supplement nicotinamide riboside (ChromaDex, Irvine CA).
  NR is distributed by ChromaDex, Inc., Irvine, CA. NR is available as 300 mg capsules.
  The dietary supplement will be re-labeled by the Hospital of the University of Pennsylvania (HUP) Investigational Drug Service according to FDA regulations, including subject and physician name and NR or Placebo 300 mg capsules.
  Arms: Exercise Intervention and NR; Nicotinamide Riboside (NR)
Dietary Supplement: Placebo — The matched placebo will contain the same excipients without the active supplement and is generally recognized as safe. The placebo will be covered in an identical capsule (NR will be covered in the same capsule)
  Arms: Exercise Intervention and Placebo; Placebo
Other: Exercise Intervention — The exercise program consists of at-home training sessions and will include aerobic and strengthening components designed to progress persons gradually to 150-300 minutes of the equivalent of moderate aerobic activity, and twice weekly strengthening over 16 weeks. For aerobic training, the eventual intensity and duration goal (adapted for each person as necessary) will be for persons to train at 70-80% of peak 2MSPT heart rate 20-45 minutes 3-5 days/week. For resistance exercises the goal will be a load/weight that results in fatigue after 3 sets of 10-12 repetitions on 8-10 exercises 2 days/week.
  Arms: Exercise Intervention and NR; Exercise Intervention and Placebo

SUMMARY:
This will be a randomized, placebo-controlled trial with a 2x2 factorial design testing the effects of an NAD+ precursor (NR) and exercise on skeletal muscle quality and VO2max in AYA HCT survivors.

The primary outcome is the change in muscle strength (isometric knee extension) from baseline to 16 weeks. Key secondary outcomes are the change in muscle strength (ankle plantarflexion) from baseline to 16 weeks, the change in grip strength from baseline to 16 weeks, the change in lower extremity muscle mass from baseline to 16 weeks, the change in muscle OXPHOS capacity from baseline to 16 weeks, and the change in aerobic capacity (VO2 max) from baseline to 16 weeks.

DETAILED DESCRIPTION:
Adolescents and young adults (AYAs) who undergo hematopoietic cell transplantation (HCT) are at an especially high risk of developing sarcopenia (loss of skeletal muscle mass), which occurs earlier than would be expected from advancing age alone. This is important as not only it doubles their risk for non-relapse mortality, but it also leads to premature cardiovascular disease. The investigators propose a mechanistic randomized controlled trial of home-based remotely supervised exercise (aerobic and resistance) training and supplementation with nicotinamide riboside, a precursor of NAD+, a metabolite that is critical for muscle metabolism, in AYA survivors of HCT. The findings will lay the critical groundwork for future trials to prevent or mitigate the myriad downstream adverse effects of low muscle mass in AYA HCT survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ages 10-30 years at enrollment
2. Able to understand and speak English
3. Diagnosis of leukemia (myeloid, lymphoid), aplastic anemia, bone marrow failure syndrome, or myelodysplastic syndrome requiring allogeneic HCT
4. 6-48 months from allogeneic HCT
5. Females must have a negative urine/serum pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
6. Subject's informed consent or parental/guardian permission (informed consent) and if appropriate, child assent
7. Minimum weight of 24 kg

Exclusion Criteria:

1. Known sensitivity to NR
2. Concurrent use of any medications, including statins, likely to increase risk of NR toxicity
3. Active malignancy, investigational agent(s) within 4 wks, or supraphysiological glucocorticoids at the baseline visit
4. Currently meeting public health exercise guidelines
5. Use of NAD+ precursors (supra-physiologic) within 4 weeks
6. Hemoglobin < 10 g/dL
7. Platelets < 50K
8. Diabetes Mellitus requiring insulin or insulin secretagogue
9. HbA1C ≥ 8% or fasting glucose > 125 mg/dL; However if the participant is diabetic, both fasting glucose level and HbA1C must meet the criteria to be deemed eligible.
10. Kidney disease (eGFR < 60 ml/min/1.73 m2)
11. Liver disease Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) (ALT/AST > 3 x ULN)
12. Limitations in physical function preventing exercise testing/training
13. Unstable angina or history of acute myocardial infarction (<5 days of planned study procedures)
14. Recurrent syncope
15. Symptomatic severe aortic stenosis
16. Uncontrolled arrhythmia causing symptoms
17. Pulmonary embolus <3 months of study procedures
18. Thrombosis of lower extremities
19. Symptomatic moderate or severe persistent asthma based on Forced Expiratory Volume (FEV) from pre-HCT pulmonary function testing
20. Room air desaturation at rest ≤85%
21. Females: Pregnant or planning pregnancy
22. Non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (e.g. infection, renal failure, thyrotoxicosis, >moderate Graft versus host disease (GVHD) resulting in physical or functional impairment)
23. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
24. For MRI procedure: Contraindications to MRI. Individuals will be screened to ensure they can safely complete the MRI. *participants who cannot complete the MRI will not be excluded from participation in the remainder of the study procedures if they meet those inclusion and exclusion criteria.
25. Current weight precludes safe completion of study procedures

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Within participant changes in muscle strength (Isometric knee extension, Z-score) | Baseline to 16 Weeks
  Muscle Strength will be assessed by completion of isometric contractions using a Biodex dynamometer.

SECONDARY OUTCOMES:
Within participant change in muscle strength (Ankle Plantarflexion) | Baseline to 16 Weeks
  Muscle Strength will be assessed by completion of isometric contractions using a Biodex dynamometer.
Within participant change in grip strength (Hand Grip Dynamometry) | Baseline to 16 Weeks
  Grip Strength will be assessed using a hand grip dynamometry device.
Within participant changes in muscle mass (lower leg lean muscle mass by DXA) | Baseline to 16 Weeks
  Muscle mass will be assessed by completion of whole body DXA scanning.
Within participant changes in post-exercise oxidative phosphorylation capacity (OXPHOS). | Baseline to 16 Weeks
  OXPHOS capacity will be assessed by completion of non-invasive MRI scanning using creatine chemical exchange saturation transfer (CrCEST).
Within participant change in aerobic capacity (VO2 max, Maximal Oxygen Uptake on Cardiopulmonary Exercise Testing). | Baseline to 16 Weeks
  VO2 Max will be assessed by completion of an incremental cardio-pulmonary Exercise Stress Test (EST) on an upright leg cycle ergometer

CONTACTS AND LOCATIONS:
Overall Officials: Sogol Mostoufi-Moab, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
No identifiable data will be used for future study without first obtaining IRB approval. The investigator will obtain a fully executed data use agreement between the provider (the PI) of the data and any recipient researchers [(including others at CHOP) before sharing a limited dataset (or the data will only be provided to users under a fully executed data use (or data sharing) agreement approved by the Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB)]. The execution of the agreement will require approval by the Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB) or a demonstration of IRB exemption per institutional policy.
Time Frame: The investigator will make data available after the completion of the trial and posting of results on ClinicalTrials.gov and in conjunction with NIH policies.
Access Criteria: Access will be limited to only using the data for research purposes that do not identify an individual participant and ensuring the data is securely maintained.

REFERENCES:
- [Derived] Song M, Armenian SH, Bhandari R, Lee K, Ness K, Putt M, Lindenfeld L, Manoukian S, Wade K, Dedio A, Guzman T, Hampton I, Lin K, Baur J, McCormack S, Mostoufi-Moab S. Exercise training and NR supplementation to improve muscle mass and fitness in adolescent and young adult hematopoietic cell transplant survivors: a randomized controlled trial 1. BMC Cancer. 2022 Jul 19;22(1):795. doi: 10.1186/s12885-022-09845-1. PMID 35854224